CLINICAL TRIAL: NCT02834026
Title: Impact of the Cycle Ergometer in Muscle Strength and Pulmonary Function in Patients in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Profa. Dra. Vera Lúcia dos Santos Alves, PHD, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1.398.846
Record Dates: First submitted 2016-07-05; First posted 2016-07-15 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Chronic Renal Disease; Renal Dialysis
Keywords: Muscle Strength; Muscle Strength Dynamometer; Chronic Renal Disease; Exercise; Physical therapy modalities
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention group held two months of training in hemodialysis a physical therapy protocol with cycle ergometer
  Interventions: Other: Cicloergometry training
- Control (Experimental): The control group was reassessed after two months of the initial evaluation
  Interventions: Other: No Cicloergometry training

INTERVENTIONS:
Other: Cicloergometry training
  Arms: Intervention
Other: No Cicloergometry training
  Arms: Control

SUMMARY:
Muscle strength can be measured by dynamometry, but the investigators did not find in the literature the study of this technique in the quadriceps of patients with chronic kidney disease on hemodialysis. Analyze training impact conducted by cycle ergometer in quadriceps muscle strength in patients with chronic kidney disease during hemodialysis. This study will be a prospective, randomized. Inclusion of 46 patients followed by the dialysis unit of a university hospital, over 18 years, of both genders who underwent hemodialysis for more than six months and signed the consent form and enlightened. Patients will be divided into two groups: Intervention (n = 23) and control (n = 23). All will be evaluated for demographics and quadriceps strength given by standardization of technique, with hard and windy belt. The control group will be reassessed after two months of the initial assessment, since the intervention group held two months of training in hemodialysis a physical therapy protocol with the cycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Performing HD over six months
* Clinically stable
* Patients no diagnosis of lung disease
* Neurological or mioarticular previous or current and agreed to participate in the study and signed informed consent and informed

Exclusion Criteria:

* Patients undergoing elective surgery or emergency six months before or during the performance of the protocol
* Cardiac decompensation
* Used continuous or nocturnal oxygen
* Patients using bracing of the lower limbs.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Muscle strength evaluated by dynamometry | Two months
  dynamometry
Peripheral blood tests | Two months
  hemoglobin (g / dL)
Peripheral blood tests | Two months
  serum albumin (GDL)
Peripheral blood tests | Two months
  Creatinine (mg / dL)
Peripheral blood tests | Two months
  Urea (mg / dL)
Peripheral blood tests | Two months
  Kt / V

CONTACTS AND LOCATIONS:
Locations (1):
- Vera Lúcia dos Santos Alves, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639